CLINICAL TRIAL: NCT04227067
Title: The Use of TENS for the Treatment of Back Pain in the Emergency Department
Brief Title: TENS for Back Pain Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Adam Singer, Professor and Vice Chairman for Research, Stony Brook University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB2019-00435
Record Dates: First submitted 2020-01-10; First posted 2020-01-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Back Pain
Keywords: TENS, back pain, ibuprofen
MeSH Terms: conditions — Back Pain | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- TENS (Active Comparator): A TENS device consists of an electric pulse generator and pads that are attached to the skin on around the area of maximal pain. We will use the conventional mode, which provides nerve stimulation with a pulse width of 60 microseconds and a pulse rate of 60 pulses per second. The channel intensity will be gradually increased until the intensity is noticeable but not painful.
  Interventions: Device: TENS
- SHAM TENS (Sham Comparator): In the SHAM TENS group the TENS pads will be attached to the pulse generator and the patients skin around the painful area. The investigator will turn the knobs on but the batteries will be removed from the device.
  Interventions: Device: SHAM TENS

INTERVENTIONS:
Device: TENS — An electrical impulse is delivered to the skin around the painful area using pads attached to an electric generator.
  Arms: TENS
Device: SHAM TENS — A TENS generator without batteries is used. The pads are attached to the generator and to the skin around the painful area.
  Arms: SHAM TENS

SUMMARY:
In this study we will see if application of TENS for a period of 30 minutes in addition to ibuprofen reduces the pain of emergency department patients with back pain compared with ibuprofen and a sham TENS unit.

DETAILED DESCRIPTION:
Adult patients presenting to the emergency department with moderate to severe back pain of relatively short duration without neurological deficits will be eligible for inclusion in the study. After signing informed consent the patients will rate their pain severity and receive a 400 mg dose of ibuprofen and then randomly be assigned to either TENS or sham TENS for 30 minutes. At the end of the study period patients will again be asked to rate their pain severity and indicate whether their pain got better or worse. We will also ask them to try and guess which treatment they received and whether they require any medications for their pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 years or greater
* Able to consent
* Back pain of less than 2 weeks duration
* Pain severity of at least 5/10 on a verbal numeric scale from 0 (none) to 10 (worst)

Exclusion Criteria:

* Pregnant patients
* Minors
* Prisoners
* Neurological deficits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2024-02-12 (Actual); Study Completion 2024-02-12 (Actual)

PRIMARY OUTCOMES:
Pain severity | 30 minutes after application of TENS unit
  Pain severity graded on a verbal numeric pain scales from none (0) to most (10)

SECONDARY OUTCOMES:
Use of rescue medications | 30 minutes after application of the TENS unit
  The percentage of patients that were administered an additional analgesic medication after the application of TENS

CONTACTS AND LOCATIONS:
Overall Officials: Adam Singer, MD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Otterness K, McMahon B, Ma M, Thode HC Jr, Singer AJ. The use of TENS for the treatment of back pain in the emergency department: A randomized controlled trial. Acad Emerg Med. 2025 Aug;32(8):828-835. doi: 10.1111/acem.70013. Epub 2025 Apr 9. PMID 40202296